CLINICAL TRIAL: NCT05220774
Title: Effectiveness, Adverse Event Rates and Patient Tolerability of ERCP With Conscious Sedation Versus Anesthesia
Brief Title: Conscious Sedation Versus Anesthesia for ERCP
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: McGill University (Other); University of Ottawa (Other); Queen's University (Other); Halton Health (Oakville) (Unknown); Island Health, Victoria, BC (Other); Radboud Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: REB21-1887
Record Dates: First submitted 2021-11-30; First posted 2022-02-02 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: ERCP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anesthetist-administered sedation (AAS): Patients undergoing ERCP and receiving AAS
- endoscopist-directed conscious sedation (EDCS): Patients undergoing ERCP and receiving EDCS

SUMMARY:
Studies directly comparing EDCS with AAS during ERCP are scarce, varying widely in their designs and reaching conflicting conclusions regarding safety and effectiveness. The investigators will assess, via a multi-center prospective study, the success, adverse event rates, and patient tolerability of ERCP when performed under AAS versus EDCS.

DETAILED DESCRIPTION:
1. Background and Rationale

   Endoscopic retrograde cholangiopancreatography (ERCP) is critical in the diagnosis and therapy of pancreatico-biliary conditions. In contrast to routine upper and lower gastrointestinal (GI) endoscopic procedures, ERCP has several unique characteristics that require consideration when formulating a sedation plan. Factors such as patient comorbidities, positioning, airway issues, and longer procedure times collectively contribute to a high risk of sedation-related adverse events (SRAEs) during ERCP.

   In contrast to the United States (US), where anesthetist-administered sedation (AAS) for ERCP is the norm, endoscopist-directed conscious sedation (EDCS) remains the primary method of sedation for ERCP in the United Kingdom (UK), Canada, and other countries with publicly funded national healthcare systems. This practice is largely driven by resource availability and cost limitations. AAS typically involves either general endotracheal anesthesia (GEA) or deep sedation without an endotracheal tube, often referred to as monitored anesthesia care (MAC).

   Studies directly comparing EDCS with AAS during ERCP are scarce, varying widely in their designs and reaching conflicting conclusions regarding safety and effectiveness. Furthermore, little is known regarding the sedation method as it relates to procedure-related adverse events (AEs). Finally, patient-reported experience measures (PREMs) in this field have been insufficiently studied to date. The heterogenous nature and inconsistent findings of existing studies comparing AAS and EDCS necessitate further study with data of higher quality and granularity.
2. Research Question and Objectives

   The investigators will assess, via a multi-center prospective study, the success, adverse event rates, and patient tolerability of ERCP when performed under AAS versus EDCS.
3. Methods

A total of 9 sites will participate using data from the Calgary Registry for Advanced and Therapeutic Endoscopy (CReATE). An anticipated 85% of procedures across included sites will be performed under EDCS, with the remainder performed under AAS. Consecutive patients ≥ 18 years of age undergoing ERCP will be included if informed consent is obtained. The investigators will collect information on 1) patient demographics and risk factors (including but not limited to Sphincter of Oddi dysfunction, prior acute or recurrent pancreatitis, and relevant medications) and 2) procedural details (including but not limited to cannulation attempts, cannulation time, trainee involvement and post-ERCP pancreatitis [PEP] prophylaxis). At the time of discharge from the endoscopy unit, outpatients will be assessed using the Patient-reported Scale for Tolerability of Endoscopic Procedures (PRO-STEP), a validated tool that measures intra- and post-procedural physical tolerability.

Thirty days after index ERCPs, research staff will contact patients using standardized interview scripts in addition to performing electronic medical record reviews to assess for any adverse events, defined using the American Society for Gastrointestinal Endoscopy (ASGE) Lexicon.

The primary outcome will be the procedural success of ERCP, defined using a previously published set of a priori criteria. Secondary outcomes will include immediate and delayed adverse event rates (including SRAEs, PEP, clinically significant bleeding, and cholangitis/sepsis), patient tolerability (as assessed by PRO-STEP), total cannulation attempts, pancreatic duct (PD) cannulation, rates of pre-cut sphincterotomy or needle-knife papillotomy (NKP), cannulation time, and overall procedure time (from esophageal intubation to extubation). SRAEs will be defined as any of the following: oxygen saturation < 85% for a sustained period of 60 seconds, requirement for mask ventilation or unplanned endotracheal intubation, intraprocedural use of one or more vasopressors or reversal agent(s), hypotension with systolic blood pressure < 90 mm Hg requiring treatment, cardiac and/or respiratory arrest, or death. PRO-STEP scores of >6 (on a scale of 0-10) will be considered to represent poor intraprocedural tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Subject referred for ERCP for biliary indication;
* Subject has not undergone prior ERCP, sphincterotomy, and/or sphincteroplasty;
* Subject age 18 years or older;
* Subject able to give informed consent to involvement be included.

Exclusion Criteria:

* Subject has a standard contraindication to ERCP;
* Subject or surrogate unable or unwilling to provide informed consent;
* Subject age < 18 years;
* Pancreatic indication for ERCP;
* Morbid obesity;
* Known history of difficult sedation and/or failed medical procedure(s), endoscopy or other, using EDCS;
* Planned cholangioscopy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred to a hospital-based endoscopy unit for consideration of ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 3174 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
procedural success of ERCP | 1 day
  Defined using a previously published set of a priori criteria by indication (Forbes et al. BMC Gastroenterology 2020; 20:64).

SECONDARY OUTCOMES:
post-ERCP pancreatitis | 30 days
  Defined using a previously published set of a priori criteria by indication (Cotton et al. Gastrointest Endoscopy 2010; 71:446-54).
post-ERCP bleeding | 30 days
  Defined using a previously published set of a priori criteria by indication (Cotton et al. Gastrointest Endoscopy 2010; 71:446-54).
post-ERCP cholangitis | 30 days
  Defined using a previously published set of a priori criteria by indication (Cotton et al. Gastrointest Endoscopy 2010; 71:446-54).
patient tolerability | 1 day
  Defined on patient-reported scale for tolerability of endoscopic procedures (PRO-STEP) - Forbes et al. Gastrointest Endosc 2021; 94: 103-10 - measured from 0 to 10 in all domains.

CONTACTS AND LOCATIONS:
Overall Officials: Nauzer Forbes, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Peter Lougheed Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Deidentified aggregate-level data may be available upon reasonable request.